CLINICAL TRIAL: NCT04911933
Title: Development of Mental Health Outcomes Following the 2020 Petrinja Earthquake in Croatia: a Longitudinal Study
Brief Title: Development of Mental Health Outcomes Following the 2020 Petrinja Earthquake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuropsychiatric Hospital dr Ivan Barbot (Other)
Responsible Party: Principal Investigator, Dragan Puljic, MD, Psychiatrist Consultant, Neuropsychiatric Hospital dr Ivan Barbot
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZH/MS/2176-128-14-688-3/21
Record Dates: First submitted 2021-03-12; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Mental Health Disorder; Post Traumatic Stress Disorder; Depression; Anxiety; Panic Disorder
Keywords: disaster; earthquake; mental health; family therapy; resilience; social support; systemic psychotherapy; narrative psychotherapy
MeSH Terms: conditions — Mental Disorders; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Panic Disorder; Psychological Well-Being | interventions — Family Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The form of treatment involve systemic family therapy sessions every two weeks about an hour each.
  Interventions: Behavioral: Family Therapy
- Waitlist Control (No Intervention): Participants assigned to the control condition will be placed on a waitlist for future enrollment. After primary data collection has ceased, those assigned to the control arm will receive the identical intervention delivered in the experimental condition.

INTERVENTIONS:
Behavioral: Family Therapy — There will be systemic family psychotherapy sessions every two weeks. Families and individuals who require a more intensive service will be referred to a higher level of care.
  Other Names: Systemic Psychotherapy; Narrative Psychotherapy; Collaborative Therapy
  Arms: Intervention

SUMMARY:
On 29 December 2020, an earthquake struck Petrinja in Croatia. The aim of this study is to assesses prevalence of symptoms of posttraumatic stress disorder, depression, anxiety, and panic disorder among exposed inhabitants and examine the effect of family therapy on mental health as part of a public health emergency response and rapid assessment.

DETAILED DESCRIPTION:
The strong earthquake measuring 6.4 on the Richter scale hit the area of Petrinja town in Croatia on December 29 2020, causing numerous casualties and widespread material damage. The maximum felt intensity was estimated at VIII (Heavily damaging) to IX (Destructive) on the European macroseismic scale, and it is the worst earthquake in Croatia in the last 140 years. Since the initial strong earthquake, the Petrinja area has been hit by numerous aftershocks, magnitudes ranging from 1.2 to 4.8 on the Richter scale, increasing distress of residents and contributing to further damage of houses and buildings. The earthquake and the constant aftershocks caused strong psychological and physiological reactions in children and adults directly affected as well as a large population of people living in the surrounding areas at the time when Croatia was facing a second "lockdown" during the COVID-19 pandemic.

As part of a public health emergency response, we conducted a rapid assessment among survivors in the most severely affected area by the earthquake. Findings from previous researches among survivors of natural disasters have been mixed in prevalence of mental health problems and treatments outcomes. The aim of this study is to assesses prevalence of symptoms of posttraumatic stress disorder, depression, anxiety, and panic disorder among exposed inhabitants and examine the effect of systemic family therapy on mental health during the first year following the earthquake. Qualitative methodology will be used to augment quantitative findings. The study sample consisted of 350 individuals residing in the earthquake area. Participants were selected from total number of patients requested psychological and psychiatric help during first two months after disaster. A follow up study will be conducted at 6 and 12 months to assess the change in their mental health status.

ELIGIBILITY:
Inclusion Criteria:

* People were in the earthquake area while it occured

Exclusion Criteria:

* People were not in the earthquake area while it occured

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Post traumatic stress symptoms - Assessing change over time | baseline, 6 months, 12 months
  Post traumatic stress disorder symptoms using PTSD Checklist for DSM-5 (PCL-5) which is 4 item self-report questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. It was was modified to make questions earthquake specific. The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely.".Higher score indicates higher symptoms for PTSD.
Depression and anxiety symptoms - Assessing change over time | baseline, 6 months, 12 months
  The Patient Health Questionnaire-4 (PHQ-4) is self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). The PHQ-4 questionnaire answered on a four point Likert-type scale as "None", "Mild", "Moderate" or "Severe". Higher score indicates higher symptoms for depression and anxiety.
Panic disorder symptoms - Assessing change over time | baseline, 6 months, 12 months
  Symptoms of panic disorder using the Severity Measure for panic disorder (PDSS), 7 item self-report questionnaire. Each item on the measure is rated on a 5-point scale (0=Never; 1=Occasionally; 2=Half of the time; 3=Most of the time, and 4=All of the time). The average total score is calculated by dividing the raw total score by number of items in the measure, with higher scores indicating greater severity of panic disorder symptoms.

SECONDARY OUTCOMES:
Resilience- Assessing change over time | baseline, 6 months, 12 months
  The six items of the Brief resilience scale (BRS) assess resilience as bouncing back from stress, whether it is related to resilience resources, and whether it is related to important health outcomes. BRS include an equal number of positive and negatively worded items. The BRS is scored by reverse coding items on scale from 1 to 5. Higher score indicates higher resilience.
Social support - Assessing change over time | baseline, 6 months, 12 months
  Oslo social support OSSS-3 consists of three items assessing the level of social support. The sum score ranges from 3 to 14, This continuous score was used to generate the normative data for the OSSS-3 for each scoring point as well as to determine group differences according to age and sex. The OSSS-3 sum score can be operationalized into three broad categories of social support. 3-8 poor social support ; 9-11 moderate social support; 12-14 strong social support

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Puljic, MD, Principal Investigator — Neuropsychiatric Hospital dr Ivan Barbot
Locations (1):
- Neuropsychiatric Hospital dr Ivan Barbot, Petrinja, Croatia

IPD SHARING:
Plan to Share IPD: No